CLINICAL TRIAL: NCT03976310
Title: Computed Tomography Air-trapping Characterisation for the Early Identification of Benralizumab Responders Among Eosinophilic Asthma Patients
Brief Title: CT Air-trapping for the Early Identification of Benralizumab Responders Among Eosinophilic Asthma Patients
Acronym: BenraliScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0016; 2018-002292-18 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2022-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: This single arm protocol will study individual patient responses to 12 months of benralizumab treatment and early means of detecting them. The model is a prognostic study that will use information detected via baseline quantitative thoracic computed tomography for predicting improvement in exacerbation rate 52 weeks after the start of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The study population (Other): The study population corresponds to severe eosinophilic asthma patients (see eligibility criteria).
  Interventions: Drug: 48 weeks of Benralizumab; Other: Computed tomography

INTERVENTIONS:
Drug: 48 weeks of Benralizumab — Benralizumab is administered for 48 weeks (week 0 to week 48) every 4 weeks for the first 3 injections (30 mg sc per injection), and then every 8 weeks for the following 5 injections.
Other: Computed tomography — Computed tomography of the thorax is performed at the beginning (week 0), middle (week 24) and towards the end (week 48) of Benralizumab therapy. A sinus scan is also added on weeks 0 and 48.

SUMMARY:
BenraliScan aims to obtain thoracic computed tomography imaging data to predict the future level of patient response to a monoclonal antibody. Because the clinical responses under study can take many months to manifest, early identification of patients most-likely to benefit from treatment and treatment rule-out for others will save considerable time for everybody involved.

The primary objective of BenraliScan is to determine the prognostic value (sensitivity, specificity, positive predictive value, negative predictive value) of air-trapping measures (Expiratory/Inspiratory ratios for Mean Lung Density (MLDe/i)) detected via quantitative thoracic computed tomography at baseline for improvement in exacerbation rate (the presence of a ≥50% reduction in baseline exacerbation rate versus the absence of a ≥50% reduction in baseline exacerbation rate) at 52 weeks among eosinophilic asthma patients treated with Benralizumab.

DETAILED DESCRIPTION:
Secondary, exploratory objectives include:

* To describe clinical improvement category sub-groups (e.g. non-responders versus strong responders) in terms of: target concomitant medication usage, symptomology, quality of life (questionnaires), exacerbation rates (and other adverse events) and lung function parameters, differential blood counts, serum club cell secretory protein (CCSP) levels, other quantitative thoracic computed tomography (QTCT) variables, sinus mucosal thickness.
* To perform exploratory, prognostic-value studies (including but not limited to prognostic variables derived from changes occurring over 24 weeks and from clustering or factor mining at baseline and 24 weeks). These exploratory studies will include (but are not necessarily limited to) estimating the sensitivity/specificity of baseline/early imaging variables (or combination thereof) for predicting clinical response variables.
* To describe the prognostic categories (e.g. predicted non-responder versus predicted responder) found in terms of: clinical improvement, target concomitant medication usage, symptomology, quality of life (questionnaires), exacerbation rates (and other adverse events) and lung function parameters, differential blood counts, serum CCSP levels, other QTCT variables, sinus mucosal thickness.
* To create a centralised image library associated with the study.
* To verify the reproducibility of the relationships found between mean lung density (upper and lower lung, inspiratory and expiratory), the fractal dimension of -850 HU segmentations, and clinical variables found during the SCANN'AIR study (NCT03102749).
* To explore the association between bronchial homothety curves (the homothety of two consecutive bronchial measurements as a function of bronchial generation) and disease severity/progression.
* To monitor patient safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and acceptance of the protocol
* The patient has given his/her informed consent and signed the consent form
* Affiliation with or beneficiary of the French national health insurance system
* Female and male patients aged 18 to 75 years (inclusively) with a history of physician-diagnosed severe asthma (according to GINA criteria) requiring treatment with high-dose inhaled corticosteroid (ICS) plus long-acting beta-agonists for at least 12 months prior to inclusion
* Documented current treatment with high daily doses of ICS (>1000 µg equivalent beclomethasone) plus at least one other asthma controller for at least 6 months prior to inclusion
* History of at least 2 asthma exacerbations while on ICS plus another asthma controller that required treatment with systemic corticosteroids (any administration route) in the 12 months prior to inclusion. For patients receiving corticosteroids as a maintenance therapy, the corticosteroid treatment for the exacerbation is defined as a temporary increase in their maintenance dose.
* Uncontrolled disease (Asthma Control Questionnaire >1.5)
* Pre bronchodilator forced expiratory volume at 1 second (% predicted) between 40% and 85%, established according to the NHANESIII criteria
* Blood eosinophilia ≥ 300 cells / µl at least once during the previous 12 months -OR- blood eosinophilia ≥ 300 cells / µl upon inclusion
* Women of childbearing potential must use at least one acceptable and effective form of birth control
* Weight ≥ 40 kg

Exclusion Criteria:

* Other respiratory diseases or associated lung infections
* Patient treated with a monoclonal antibody in the 5 months preceding inclusion
* Patient who participated in a therapeutic study in the month prior to inclusion
* Patient deprived of liberty by judicial or administrative decision
* Major (adult) protected by the law (under any kind of guardianship)
* Patient in an exclusion period determined by another protocol
* Patient who participated in another research protocol with X-ray exposure in the past 12 months
* Patient who has already participated in the present protocol
* Hypersensitivity to benralizumab or to any of the excipients: histidine, histidine hydrochloride monohydrate, trehalose dehydrate, polysorbate 20 and water for injections
* Exacerbation, antibiotics, or non-maintenance systemic steroids during the 6 weeks prior to inclusion
* Subjects with untreated helminthic parasitic infection
* Lactating or pregnant* females or females who intend to become pregnant
* Subjects with a history of anaphylaxis to any biologic therapy
* Subjects taking immunosuppressive medications (except oral prednisone and inhaled and topical corticosteroids)
* Subjects with intercurrent illnesses (eg, viral illnesses) that may compromise the safety of the subject
* Subjects who are febrile (≥ 38°C)
* Currently smoking or smoking history ≥ 20 pack years
* Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date of informed consent, and assent when applicable was obtained
* Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date of informed consent, and assent when applicable, was obtained

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
The prognositc value (sensitivity) of baseline expiratory to inspiratory mean lung density (MLDe/i) for predicting improvement in exacerbation rate | 52 weeks
  The sensitivity and specificity of the baseline expiratory to inspiratory mean lung density (MLDe/i) for predicting improvement in exacerbation rate (the presence of a ≥50% reduction in baseline exacerbation rate versus the absence of a ≥50% reduction in baseline exacerbation rate) at week 52.
The prognositc value (specificity) of baseline expiratory to inspiratory mean lung density (MLDe/i) for predicting improvement in exacerbation rate | 52 weeks
  The sensitivity and specificity of the baseline expiratory to inspiratory mean lung density (MLDe/i) for predicting improvement in exacerbation rate (the presence of a ≥50% reduction in baseline exacerbation rate versus the absence of a ≥50% reduction in baseline exacerbation rate) at week 52.

SECONDARY OUTCOMES:
52E: the number of exacerbations occurring during follow-up | 52 weeks
  An exacerbation is defined as follows: worsening of symptoms (increased shortness of breath, cough, sputum, with or without fever) which necessitates unscheduled healthcare resource use, a need for >48h of oral corticosteroids. For oral steroids, a minimal dose of 0.25 mg/kg is required. For patients taking oral steroids on a long term basis, at least a doubling dose for 2 days is required.
52cFEV1 pre BD: The change in forced expiratory volume in 1 second (FEV1) pre BD from baseline | 52 weeks
52cACQ: The change from baseline in the ACQ score | 52 weeks
  'ACQ' refers to the Asthma Control Questionnaire: The ACQ-6 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
52CI: A clinical improvement score | 52 weeks
  52CI: A clinical improvement score starting at zero and where points are added based on the following criteria:
  * 52E = 0 or 1 non-admitting† exacerbation (+1 point);
  * 52cFEV1 pre BD > 300 ml in asthma patients (+1 point);
  * 52cACQ > 0.5 (+1 point).
Concomitant medication use | 52 weeks
The Asthma Control Questionnaire | Week 0
  'ACQ' refers to the Asthma Control Questionnaire: The ACQ-6 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
The Asthma Control Questionnaire | Week 24
  'ACQ' refers to the Asthma Control Questionnaire: The ACQ-6 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
The Asthma Control Questionnaire | Week 52
  'ACQ' refers to the Asthma Control Questionnaire: The ACQ-6 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
The SNOT22 Questionnaire | Week 0
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
The SNOT22 Questionnaire | Week 24
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
The SNOT22 Questionnaire | Week 52
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
The Asthma Quality of Life Questionnaire (AQLQ) | Week 0
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain questionnaire with a 2-week recall period. Each item is scored using a 7-point likert scale where scores range from 1 to 7 and higher scores indicate higher quality of life. Simple means are used to calculate the overall AQLQ score (as well as domain scores).
The Asthma Quality of Life Questionnaire (AQLQ) | Week 24
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain questionnaire with a 2-week recall period. Each item is scored using a 7-point likert scale where scores range from 1 to 7 and higher scores indicate higher quality of life. Simple means are used to calculate the overall AQLQ score (as well as domain scores).
The Asthma Quality of Life Questionnaire (AQLQ) | Week 52
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain questionnaire with a 2-week recall period. Each item is scored using a 7-point likert scale where scores range from 1 to 7 and higher scores indicate higher quality of life. Simple means are used to calculate the overall AQLQ score (as well as domain scores).
Functional residual lung capacity | Week 0
Functional residual lung capacity | Week 52
Residual lung volume | Week 0
Residual lung volume | Week 52
The ratio of residual volume over total lung capacity | Week 0
The ratio of residual volume over total lung capacity | Week 52
Pre-bronchodilator forced expiratory volume in 1 second (litres) | Week 0
Pre-bronchodilator forced expiratory volume in 1 second (litres) | Week 24
Pre-bronchodilator forced expiratory volume in 1 second (litres) | Week 52
Pre-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 0
Pre-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 24
Pre-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 52
Pre-bronchodilator forced vital capacity (litres) | Week 0
Pre-bronchodilator forced vital capacity (litres) | Week 24
Pre-bronchodilator forced vital capacity (litres) | Week 52
Pre-bronchodilator forced vital capacity (% predicted) | Week 0
Pre-bronchodilator forced vital capacity (% predicted) | Week 24
Pre-bronchodilator forced vital capacity (% predicted) | Week 52
Pre-bronchodilator forced expiratory volume in 1 second / forced vital capacity | Week 0
Pre-bronchodilator forced expiratory volume in 1 second / forced vital capacity | Week 24
Pre-bronchodilator forced expiratory volume in 1 second / forced vital capacity | Week 52
Post-bronchodilator forced expiratory volume in 1 second (litres) | Week 0
Post-bronchodilator forced expiratory volume in 1 second (litres) | Week 24
Post-bronchodilator forced expiratory volume in 1 second (litres) | Week 52
Post-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 0
Post-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 24
Post-bronchodilator forced expiratory volume in 1 second (% predicted) | Week 52
Complete blood count | Week 0
Complete blood count | Week 24
Complete blood count | Week 52
Club cell secretory protein (CCSP) (ng / ml) | Week 0
Club cell secretory protein (CCSP) (ng / ml) | Week 52
The ratio of expiratory to inspiratory mean lung density | Week 0
The ratio of expiratory to inspiratory mean lung density | Week 24
The ratio of expiratory to inspiratory mean lung density | Week 48
LAA-850: The % lung attenuation area at -850 hounsfield units | Week 0
LAA-850: The % lung attenuation area at -850 hounsfield units | Week 24
LAA-850: The % lung attenuation area at -850 hounsfield units | Week 48
The fractal dimension of LAA-850 | Week 0
The fractal dimension of LAA-850 | Week 24
The fractal dimension of LAA-850 | Week 48
LAA-950: The % lung attenuation area at -950 hounsfield units | Week 0
LAA-950: The % lung attenuation area at -950 hounsfield units | Week 24
LAA-950: The % lung attenuation area at -950 hounsfield units | Week 48
The fractal dimension of LAA-950 | Week 0
The fractal dimension of LAA-950 | Week 24
The fractal dimension of LAA-950 | Week 48
Normalized bronchial parietal thickness | Week 0
  From bronchial morphometry characterization on computed tomography scan
Normalized bronchial parietal thickness | Week 24
  From bronchial morphometry characterization on computed tomography scan
Normalized bronchial parietal thickness | Week 48
  From bronchial morphometry characterization on computed tomography scan
Thickness of the sinus mucosa | Week 0
Thickness of the sinus mucosa | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Bommart, MD PhD, Study Director — University Hospitals of Montpellier, France
Locations (2):
- France (2):
  - Assistance Publique - Hopitaux de Marseille, Marseille
  - University Hospitals of Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No